CLINICAL TRIAL: NCT06967090
Title: Accuracy of Guided Implant Placement Using Artificial Intelligence Segmentation Versus Conventional Technique: A Randomized Clinical Trial
Brief Title: Accuracy of Guided Implant Placement Using Artificial Intelligence Segmentation Versus Conventional Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Dina Emad Rabie, Principal Investigator, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI in Guided implant surgery
Record Dates: First submitted 2025-05-01; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Dental Implant
Keywords: AI in guided dental implant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: (Active Comparator): Will use surgical guided implant using AI tooth segmentation of the CBCT alone without intraoral scan to fabricate the implant guide.
  Interventions: Device: Implant surgery using surgical guide
- Control group: (Active Comparator): Will use surgical guided implant using conventional technique and intraoral scan to fabricate the implant guide.
  Interventions: Device: Implant surgery using surgical guide

INTERVENTIONS:
Device: Implant surgery using surgical guide — Dental implant surgical guides are customized device used to position dental implants to ensure that the implant is placed in the most ideal location, angulation and depth into the bone.

SUMMARY:
To compare the accuracy of surgical guided implant using AI tooth segmentation of the CBCT alone without intraoral scan to fabricate the implant guide versus conventional technique by alignment the CBCT and intraoral scan to fabricate the implant guide in posterior implant.

DETAILED DESCRIPTION:
Background:

Implant dentistry has developed rapidly all around the world in the past few decades. A revolutionary change in the field of implant dentistry has been brought forward by Artificial intelligence (AI) technology. Many advantages come from the use of guided implant surgery and virtual implant planning, including optimal surgical and prosthetic treatment plan and predictable and effective application.

Statement of the problem:

Even with over ten years of clinical and research data, as well as advancements in apparatus and technique, there are still discrepancies between planned and achieved implant placements when using conventional guided implant surgery.

Review of literature:

Conventional guided implant surgery is considered the gold standard for implant placement as it provides a higher degree of accuracy and a lower risk of complications after surgery. Conventional guided implant surgery consists of 3 key steps. The first step is obtaining a 3D model of the manually segmented CBCT and a 3D model of the intraoral scan (IOS). The second step is alignment of the 3D model of the CBCT and the IOS by Iterative Closest Point Alignment (ICP Alignment). The third step is the virtual implant planning and surgical guide design. The segmentation is needed to create a 3D surface model from a CBCT or CT. Because of this, any error or inaccuracy in the segmentation or alignment process will lower the associated quality of virtual surgical planning.

Segmentation based on AI shows promise and saves time. This revolutionary AI-driven tool allows for precise and quick segmentation of the CBCT images. Therefore, all the steps of the conventional technique to fabricate an implant surgical guide can be less sophisticated if we use the AI segmentation alone without IOS.

Using AI tooth segmentation of the CBCT to obtain a 3D model and immediately, in one step, start virtual implant planning and designing a tooth-supported surgical guide without intraoral scan can minimize the clinical workload while opening the door for possible uses regarding digital workflows.

The outcomes of this investigation may contribute to the enhancement of pre-operative planning processes, including implant positioning and bone grafting. Still, not much has been discovered about how different segmentation techniques may affect clinical practice.

According to our knowledge there is deficiency in the literature in the evaluation of the accuracy of the AI segmentation of the CBCT when used alone in surgical implant guide without the use of intraoral scan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with missing posterior teeth require implant surgery.
2. Patients have remaining teeth that can support the surgical guide.
3. The edentulous area should involve healed bone sites at least 3 months after extraction.
4. The edentulous area should have bone height of at least 10 mm from the alveolar crest to the nearest vital structure and bone width of at least 6 mm.
5. Age: patient above 18 years old.
6. All patients are in good health with no systemic, immunologic or debilitating diseases that could affect normal bone healing.
7. All selected patients are non-smokers and non-alcoholics. Patients are free from temporomandibular disorders and abnormal (TMD) oral habits such as bruxism.

Exclusion Criteria:

1. Systemic disease that may affect bone quality.
2. Patients with poor oral hygiene and active periodontal diseases.
3. Patient with limited mouth opening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the placed implants | one week after surgery
  The accuracy of the placed implants by measurements of the following:
  Horizontal platform deviation, (Measuring unit in millimeter) corresponding to the horizontal distance between the virtually planned and actually placed implant platforms.
Horizontal apex deviation, (Measuring unit in millimeter) | one week after surgery
  corresponding to the horizontal distance between the virtually planned and placed implant apices.
Angular deviation, (Measuring unit in degree) | one week after surgery
  corresponding to the angle between the virtually planned and placed implant axes.

CONTACTS AND LOCATIONS:
Overall Officials: Haytham Ahmed Salah Al-Mahalawy, Phd, Study Chair — Head of the Department of Oral & Maxillofacial Surgery Faculty of Dentistry Fayoum University; Nourhan Mohamed Abdelmoneim, Phd, Study Chair — Lecturer of Oral & Maxillofacial Surgery Faculty of Dentistry Fayoum University

REFERENCES:
- [Background] On SW, Cho SW, Park SY, Yi SM, Park IY, Byun SH, Kim JC, Yang BE. Advancements in computer-assisted orthognathic surgery: A comprehensive review and clinical application in South Korea. J Dent. 2024 Jul;146:105061. doi: 10.1016/j.jdent.2024.105061. Epub 2024 May 9. PMID 38729289
- [Background] Altalhi AM, Alharbi FS, Alhodaithy MA, Almarshedy BS, Al-Saaib MY, Al Jfshar RM, Aljohani AS, Alshareef AH, Muhayya M, Al-Harbi NH. The Impact of Artificial Intelligence on Dental Implantology: A Narrative Review. Cureus. 2023 Oct 30;15(10):e47941. doi: 10.7759/cureus.47941. eCollection 2023 Oct. PMID 38034167
- [Background] Schubert O, Schweiger J, Stimmelmayr M, Nold E, Guth JF. Digital implant planning and guided implant surgery - workflow and reliability. Br Dent J. 2019 Jan 25;226(2):101-108. doi: 10.1038/sj.bdj.2019.44. PMID 30679852
- [Background] Mahardawi B, Jiaranuchart S, Arunjaroensuk S, Dhanesuan K, Mattheos N, Pimkhaokham A. The Accuracy of Dental Implant Placement With Different Methods of Computer-Assisted Implant Surgery: A Network Meta-Analysis of Clinical Studies. Clin Oral Implants Res. 2025 Jan;36(1):1-16. doi: 10.1111/clr.14357. Epub 2024 Sep 10. PMID 39254507
- [Background] Aghaloo T, Hadaya D, Schoenbaum TR, Pratt L, Favagehi M. Guided and Navigation Implant Surgery: A Systematic Review. Int J Oral Maxillofac Implants. 2023 May-Jun;38(suppl):7-15. doi: 10.11607/jomi.10465. PMID 37436945
- [Background] Ulbrich M, Van den Bosch V, Bonsch A, Gruber LJ, Ooms M, Melchior C, Motmaen I, Wilpert C, Rashad A, Kuhlen TW, Holzle F, Puladi B. Advantages of a Training Course for Surgical Planning in Virtual Reality for Oral and Maxillofacial Surgery: Crossover Study. JMIR Serious Games. 2023 Jan 19;11:e40541. doi: 10.2196/40541. PMID 36656632
- [Background] Marei HF, Abdel-Hady A, Al-Khalifa K, Al-Mahalawy H. Influence of surgeon experience on the accuracy of implant placement via a partially computer-guided surgical protocol. Int J Oral Maxillofac Implants. 2019 September/October;34(5):1177-1183. doi: 10.11607/jomi.7480. Epub 2019 Apr 1. PMID 30934035
- [Background] Khaohoen A, Powcharoen W, Sornsuwan T, Chaijareenont P, Rungsiyakull C, Rungsiyakull P. Accuracy of implant placement with computer-aided static, dynamic, and robot-assisted surgery: a systematic review and meta-analysis of clinical trials. BMC Oral Health. 2024 Mar 21;24(1):359. doi: 10.1186/s12903-024-04033-y. PMID 38509530
- [Background] Custodio ALN, Chrcanovic BR, Cameron A, Bakr M, Reher P. Accuracy evaluation of 3D-printed guide-assisted flapless micro-osteoperforations in the anterior mandible. Int J Comput Dent. 2022 Nov 25;25(4):387-396. doi: 10.3290/j.ijcd.b2599841. PMID 35072427
- [Background] Li Y, Lyu J, Cao X, Zhou Y, Tan J, Liu X. Accuracy of a calibration method based on cone beam computed tomography and intraoral scanner data registration for robot-assisted implant placement: An in vitro study. J Prosthet Dent. 2024 Dec;132(6):1309.e1-1309.e9. doi: 10.1016/j.prosdent.2024.08.009. Epub 2024 Sep 7. PMID 39245604
- [Background] Minnema J, Ernst A, van Eijnatten M, Pauwels R, Forouzanfar T, Batenburg KJ, Wolff J. A review on the application of deep learning for CT reconstruction, bone segmentation and surgical planning in oral and maxillofacial surgery. Dentomaxillofac Radiol. 2022 Sep 1;51(7):20210437. doi: 10.1259/dmfr.20210437. Epub 2022 May 23. PMID 35532946
- [Background] Lahoud P, Diels S, Niclaes L, Van Aelst S, Willems H, Van Gerven A, Quirynen M, Jacobs R. Development and validation of a novel artificial intelligence driven tool for accurate mandibular canal segmentation on CBCT. J Dent. 2022 Jan;116:103891. doi: 10.1016/j.jdent.2021.103891. Epub 2021 Nov 13. PMID 34780873
- [Background] Shaheen E, Leite A, Alqahtani KA, Smolders A, Van Gerven A, Willems H, Jacobs R. A novel deep learning system for multi-class tooth segmentation and classification on cone beam computed tomography. A validation study. J Dent. 2021 Dec;115:103865. doi: 10.1016/j.jdent.2021.103865. Epub 2021 Oct 26. PMID 34710545